CLINICAL TRIAL: NCT07197099
Title: Evaluation of Therapeutic Plasma Exchange for Immune-Mediated Neurological Diseases in a Sample of Egyptian Patients: An Experience at Al-Azhar University Hospitals
Brief Title: Evaluation for Therapeutic Plasma Exchange for Immune Mediated Neurological Disease
Acronym: TPE
Status: Recruiting | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Wajdi Hamid Miftah Eisay, resident, Al-Azhar University
Other Study IDs: 000110
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Neurological Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to Evaluation of Therapeutic Plasma Exchange for Immune-Mediated Neurological Diseases in a Sample of Egyptian Patients: An Experience at Al-Azhar University Hospitals, including evaluating clinical response rates and functional improvement.

DETAILED DESCRIPTION:
Therapeutic plasma exchange (TPE) is recommended as Class I therapies by the American Society for Apheresis (ASFA) guidelines and are widely used as first-line therapies for the treatment of acute neuroimmune diseases , TPE is generally well tolerated, with minor complications occurring in about 20-30% of patients ,(ASFA) publishes regular guidelines on the indications for TPE. Studies performed over the last three decades showed that myasthenia gravis (MG), Guillain-Barre syndromé (GBS) and chronic inflammatory demyelinating polyneuropathy (CIDP) were the most frequently cited indications for TPE followed by multiple sclerosis (MS) , The aims of this research to evaluate therapeutic plasma exchange for immune-mediated neurological diseases in a sample of Egyptian patients, including evaluating clinical response rates and functional improvement

ELIGIBILITY:
Inclusion Criteria:

* 1. All neurological patients irrespective of age who will undergo TPE. 2.All new and relapse cases that meet the ASFA guidelines and where TPE is the first and/or second line of therapy

Exclusion Criteria:

* 1. Individuals with contraindications to therapeutic plasma exchange, such as hemodynamic unstable, hypocalcaemia, allergy to fresh frozen plasma or albumin.

  2.Patients who will undergo fewer than five cycles of TPE and not complete the procedure.

  3.Patients with non-neurological disorders.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An Experience at Al-Azhar University Hospitals (Al-Hussein & Sayed Galal) in Egypt
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | will be conducted on each patient on two occasions: prior to and one month subsequent to the completion of plasmapheresis.
  The mRS will be rated as follows: 0, no symptoms; 1, no substantial disability; 2, slight disability; 3, moderate disability; 4, moderately severe disability; 5, severe disability; and 6, deceased.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided